CLINICAL TRIAL: NCT01391403
Title: A Double-Blind, Randomized, Placebo-Controlled Trial of Artemisinin as an Add-on Therapy to Risperidone in the Treatment of Drug-Naive First-Episode Patients With Schizophrenia
Brief Title: Artemisinin With Risperidone for First-Episode and Drug-Naive Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing HuiLongGuan Hospital (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Xiang Yang Zhang, Director, the Research Center, Beijing HuiLongGuan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMRI 05T-726
Record Dates: First submitted 2011-07-07; First posted 2011-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Risperidone; Artemisinin; Toxoplasma; Immune
MeSH Terms: conditions — Schizophrenia | interventions — artemisinin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Artemisinin, anti-toxoplasma (Experimental): Artemisinin
  Interventions: Drug: Artemisinin
- Placebo (Placebo Comparator): Placebo looks like the active drug, with the same dose.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Artemisinin — 400 mg/day
  Other Names: Qinghaosu
  Arms: Artemisinin, anti-toxoplasma
Other: Placebo — 400mg/day
  Arms: Placebo

SUMMARY:
This study will determine the effectiveness of artemisinin plus risperidone in improving symptoms and cognitive disturbances and in Chinese people with schizophrenia. The study addresses the Toxoplasma infection hypothesis of schizophrenia.

DETAILED DESCRIPTION:
Evidences of high levels of Toxoplasma gondii antibodies in the serum and the cerebrospinal fluid (CSF) of individuals with schizophrenia have suggested that this organism might be involved in the etiopathogenesis of schizophrenia. The investigators hypothesize that antimicrobial therapy by using an add-on agent together with a well-proven neuroleptic may have favorable effects on a subgroup of schizophrenic patients.

ELIGIBILITY:
Inclusion Criteria:

* Currently resides in Beijing, China
* Diagnosis of schizophrenia or schizophreniform disorder
* Duration of symptoms is no longer than 60 months
* No history of treatment with antipsychotic medication or, if previously treated, a total lifetime usage of less than 14 days
* Current psychotic symptoms are of moderate severity or greater as measured by one of the five psychotic items in the Brief Psychiatric Rating Scale (BPRS)

Exclusion Criteria:

* DSM-IV Axis I diagnosis other than schizophrenia or schizophreniform psychosis
* Documented disease of the central nervous system that might interfere with the trial assessments (e.g., stroke, tumor, Parkinson's disease, Huntington's disease, seizure disorder, history of brain trauma resulting in significant impairment, chronic infection)
* Acute, unstable, and/or significant and untreated medical illness (e.g., infection, unstable diabetes, uncontrolled hypertension)
* A clinically significant echocardiogram (ECG) abnormality in the opinion of the investigator
* Pregnant or breastfeeding
* Use of prohibited concomitant therapy
* History of severe allergy or hypersensitivity
* Dependence on alcohol or illegal drugs
* Use of any of the following medications during the trial: antipsychotic medications other than risperidone; psychostimulants; or antidepressants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2008-09; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
the Positive and Negative Syndrome Scale (PANSS) | 10 weeks

SECONDARY OUTCOMES:
the Clinical Global Impression (ICG) | 10 weeks
UKU Side Effect Rating Scale | 10 weeks
the Simpson-Angus Scale for extrapyramidal side effects (SAS) | 10 weeks
The Abnormal Involuntary Movement Scale (AIMS) | 10 weeks
the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lian Y Cao, MD, Study Chair — Beijing HuiLongGuan Hospital
Locations (1):
- Beijing HuiLongGuan hospital, Beijing, China

REFERENCES:
- See also: The Stanley Medical Research Institute (SMRI) is a nonprofit organization supporting research on the causes of, and treatments for, schizophrenia and bipolar disorder. This current study was supported by the SMRI. — http://www.stanleyresearch.org